CLINICAL TRIAL: NCT06822374
Title: Use of a Buffered 2% Hypertonic Saline Solution During Posterior Spinal Fusion
Brief Title: Hypertonic Saline in Posterior Spinal Fusion
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No funding
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chief, Department of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005116
Record Dates: First submitted 2025-01-31; First posted 2025-02-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Scoliosis Idiopathic; Scoliosis;Congenital
Keywords: intraoperative fluid resuscitation
MeSH Terms: interventions — Plasmalyte A; Ampholyte Mixtures; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypertonic saline (Experimental): Buffered 2% saline solution instead of standard of care isotonic fluid for fluid resuscitation during intraoperative care.
  Interventions: Drug: buffered 2% hypertonic saline
- Normosol-R (Active Comparator): Isotonic solution of balanced electrolytes in water for fluid resuscitation during intraoperative care.
  Interventions: Drug: Normosol-R

INTERVENTIONS:
Drug: Normosol-R — Standard of care isotonic fluid.
  Arms: Normosol-R
Drug: buffered 2% hypertonic saline — A solution containing 2% sodium chloride (NaCl) that is "buffered" by the addition of another salt like sodium acetate.
  Arms: Hypertonic saline

SUMMARY:
This is a prospective, randomized study in patients greater than or equal to 10 years of age scheduled for an posterior spinal fusion that requires invasive monitoring of arterial blood pressure. Subjects will be randomized to receive either standard of care Normosol-R or buffered 2% hypertonic saline for intraoperative fluid resuscitation.

The primary objective of this study is to compare intraoperative changes in acid-base status and electrolytes based on the type of fluid administered intraoperatively.

The secondary objective is to compare the volume of fluid required and use of adjunctive volume resuscitation with 5% albumin for intraoperative resuscitation when using standard Normosol-R or a novel buffered 2% saline solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 10 years of age
* ASA 1-3
* Undergoing a PSF procedure requiring two peripheral intravenous infusions and an arterial cannula

Exclusion Criteria:

* Arterial cannula is not indicated for the surgical procedure
* Two peripheral intravenous cannulas are not required
* An invasive arterial cannula cannot be placed

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
pH | Every 1-2 hours during the surgery
  pH level from arterial blood gas.
Base deficit | Every 1-2 hours during the surgery
  Base deficit level from arterial blood gas.
Sodium | Every 1-2 hours during the surgery
  Sodium level from arterial blood gas.
Ionized calcium | Every 1-2 hours during the surgery
  Ionized calcium level from arterial blood gas.
Potassium | Every 1-2 hours during the surgery
  Potassium level from arterial blood gas.

SECONDARY OUTCOMES:
Fluid volume | Duration of surgery (approx. 4-6 hrs.)
  Volume of fluid required for intraoperative resuscitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No